CLINICAL TRIAL: NCT05761457
Title: Efficacy and Safety of Autologous Cryopreserved Platelets in Patients With Platelet Refractoriness
Brief Title: Efficacy and Safety of Autologous Cryopreserved Platelets in Patients With PTR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20221108091732885
Record Dates: First submitted 2023-01-28; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-01

CONDITIONS: Platelet Transfusion Refractoriness
Keywords: cryopreserved autologous platelet

STUDY DESIGN:
Intervention Model Description: Prospective, single arm and multicenter study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Patients receive cryopreserved autologous platelet transfusion
  Interventions: Other: Cryopreserved autologous platelet transfusion

INTERVENTIONS:
Other: Cryopreserved autologous platelet transfusion — Autologous PLTs were collected and transfused as an individualized treatment approach, when the platelet is less than 20*10E9/L or severe bleeding occurred.

SUMMARY:
The purpose of this study is to improve the platelet level of PTR patients; Prevent and improve bleeding; Help patients to successfully through the bone marrow suppression period after chemotherapy; Reduce the overall rate of PTR and allo-immunity; Saving platelet resources and reducing blood burden.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ALL，AML，MDS, CML,CLL that suffered from PTR before, with or without HLA antibodies
* The platelet level >150*10E9/L when considering autologous PLT collection
* Age less than 70 years
* The expected life more than 3 months
* Agree to receive autologous platelet cryopreservation and infusion treatment, and sign the informed consent form

Exclusion Criteria:

* Blast cells are found in peripheral blood or bone marrow
* Patients with bacteremia or sepsis
* Coagulation function abnormality
* Patients who have a history of thrombosis and are receiving anticoagulant treatment
* Severe bleeding within 2 weeks
* Participate in another clinical study within 1 month, and have treatment with potential impact on platelets
* Patients with mental disease

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
The CCI value of 1h and 24h after cryopreserved autologous platelet transfusion | 1 hour after transfusion
  Platelet level detection
The CCI value of 1h and 24h after cryopreserved autologous platelet transfusion | 24 hours after transfusion
  Platelet level detection
The frequency or number of effective infusions (1h CCI>7.5, 24h CCI>4.5) | 1 hour after transfusion
  Corrected count increment，CCI
The frequency or number of effective infusions (1h CCI>7.5, 24h CCI>4.5) | 24 hours after transfusion
  Corrected count increment，CCI
The total platelet transfusion volume | 1 month
Incidence of adverse events after blood transfusion | 1 hour

SECONDARY OUTCOMES:
Time of platelet recovery after chemotherapy | 1 month
The overall incidence of PTR | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yue Han, PhD,MD, Principal Investigator — First Affiliated Hospital of Soochow University
Locations (1):
- First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cid J. Autologous cryopreserved platelets to overcome immune platelet refractoriness. Transfusion. 2016 Oct;56(10):2403-2404. doi: 10.1111/trf.13758. No abstract available. PMID 27739150
- [Background] Funke I, Wiesneth M, Koerner K, Cardoso M, Seifried E, Kubanek B, Heimpel H. Autologous platelet transfusion in alloimmunized patients with acute leukemia. Ann Hematol. 1995 Oct;71(4):169-73. doi: 10.1007/BF01910313. PMID 7578522
- [Background] Schiffer CA, Aisner J, Wiernik PH. Frozen autologous platelet transfusion for patients with leukemia. N Engl J Med. 1978 Jul 6;299(1):7-12. doi: 10.1056/NEJM197807062990102. PMID 661855